CLINICAL TRIAL: NCT02688985
Title: An Open-Label, Multicenter, Biomarker Study to Explore the Mechanism of Action of Ocrelizumab and B-Cell Biology in Patients With Relapsing Multiple Sclerosis or Primary Progressive Multiple Sclerosis
Brief Title: Study to Explore the Mechanism of Action of Ocrelizumab and B-Cell Biology in Participants With Relapsing Multiple Sclerosis (RMS) or Primary Progressive Multiple Sclerosis (PPMS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML29966; 2015-004616-37 (EudraCT Number)
Record Dates: First submitted 2016-02-18; First posted 2016-02-23 (Estimated); Results first posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Relapsing Multiple Sclerorsis; Multiple Sclerosis, Primary Progressive
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — ocrelizumab; Spinal Puncture; Histamine Antagonists

ARMS (5):
- RMS Cohort Arm 1: Ocrelizumab + LP (Experimental): Participants with RMS will receive ocrelizumab as two 300-mg IV infusion on Days 1 and 15 then as single infusion of 600 mg on Weeks 24 and 48. Participants will receive a LP before the start of dosing (Week 1, treatment baseline) with ocrelizumab and a second LP at Week 12. Participants will be asked to have an additional optional LP at Week 52. Participants that complete the study and continue to receive ocrelizumab will receive single infusions every 24 weeks starting from Week 72.
  Interventions: Drug: Ocrelizumab; Procedure: Lumbar Puncture; Drug: Methyloprednisolone; Drug: Antihistamine
- RMS Cohort Arm 2: Ocrelizumab + LP (Experimental): Participants with RMS will receive ocrelizumab as two 300-mg IV infusion on Days 1 and 15 then as single infusion of 600 mg on Weeks 24 and 48. Participants will receive a LP before the start of dosing (Week 1, treatment baseline) with ocrelizumab and a second LP at Week 24. Participants will be asked to have an additional optional LP at Week 52. Participants that complete the study and continue to receive ocrelizumab will receive single infusions every 24 weeks starting from Week 72.
  Interventions: Drug: Ocrelizumab; Procedure: Lumbar Puncture; Drug: Methyloprednisolone; Drug: Antihistamine
- RMS Cohort Arm 3: Ocrelizumab + LP (Experimental): Participants with RMS will receive ocrelizumab as two 300-mg IV infusion on Days 1 and 15 then as single infusion of 600 mg on Weeks 24 and 48. Participants will receive a LP before the start of dosing (Week 1, treatment baseline) with ocrelizumab and a second LP at Week 52. Participants that complete the study and continue to receive ocrelizumab will receive single infusions every 24 weeks starting from Week 72.
  Interventions: Drug: Ocrelizumab; Procedure: Lumbar Puncture; Drug: Methyloprednisolone; Drug: Antihistamine
- RMS Cohort Arm 4: Ocrelizumab + LP (Experimental): Ocrelizumab treatment will be delayed for 12 weeks from pre-treatment baseline. Participants with RMS will receive ocrelizumab as two 300-mg IV infusion on Days 1 and 15 then as single infusion of 600 mg on Weeks 24 and 48. Participants will receive a LP at Week -12 (pre-treatment baseline) and a second LP before the start of dosing (Week 1, treatment baseline). Participants will be asked to have an additional optional LP at Week 52. Participants that complete the study and continue to receive ocrelizumab will receive single infusions every 24 weeks starting from Week 72.
  Interventions: Drug: Ocrelizumab; Procedure: Lumbar Puncture; Drug: Methyloprednisolone; Drug: Antihistamine
- PPMS Cohort: Ocrelizumab + LP (Experimental): For the PPMS cohort, ocrelizumab will be administered as two 300-mg IV infusions separated by 14 days at a scheduled interval of every 24 weeks during the treatment period and then as a single 600-mg dose every 24 weeks starting week 72 during the Long-Term Extension period.
  Interventions: Drug: Ocrelizumab; Procedure: Lumbar Puncture; Drug: Methyloprednisolone; Drug: Antihistamine

INTERVENTIONS:
Drug: Ocrelizumab — Ocrelizumab will be administered as IV infusion.
  Other Names: RO4964913
Procedure: Lumbar Puncture — Participants will receive LP as specified in individual arms. Lumbar puncture is optional at week 52, except for RMS Cohort Arm 3 and PPMS Cohort. In addition, the lumbar punctures in the Long Term Extension phase is every other year.
Drug: Methyloprednisolone — Participants will receive 100 mg of IV methylprenisolone (or an equivalent) prior to ocrelizumab infusion.
Drug: Antihistamine — Participants will receive an antihistamine, such as diphenhydramine, prior to ocrelizumab infusion.

SUMMARY:
This is an open-label, multicenter, biomarker study designed to be hypothesis-generating in order to better understand the mechanism of action of ocrelizumab and B-cell biology in RMS or PPMS. The study will be conducted in two cohorts i.e. RMS cohort (4 arm group) and PPMS cohort (one arm group). RMS cohort: Ocrelizumab will be administered as two intravenous (IV) infusions of 300 milligrams (mg) on Days 1 and 15. Subsequent doses will be given as single 600-mg infusions at Weeks 24 and 48. Participants will be randomized in 1:1:1 ratio to receive lumbar puncture (LP) post-treatment at Week 12, 24, or 52 following the first dose of ocrelizumab in three arm groups. A fourth RMS arm with delayed treatment start (Arm 4 [control group]) will not be a part of the randomization and will be recruited separately, wherein treatment with ocrelizumab will be delayed for 12 weeks from pre-treatment baseline. PPMS cohort: Ocrelizumab 600 mg will be administered as two 300-mg IV infusions separated by 14 days at a scheduled interval of every 24 weeks. Participants will receive a LP at the start of the study before dosing with ocrelizumab and second LP at Week 52 following the first dose of ocrelizumab. A long-term extension will be conducted for participants that complete the study and continue to receive ocrelizumab. Treatment with ocrelizumab in the entire study will continue for approximately 4.5 years after the first infusion.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of <1 percent (%) per year during the treatment period and for at least 24 weeks after the last dose of study treatment or until their B-cells have repleted, whichever is longer

Inclusion Criteria Specific to RMS Participants:

* Diagnosis of RMS in accordance with the 2010 revised McDonald criteria
* Expanded Disability Status Scale (EDSS) score of 0 to 5.5 points, inclusive, at Screening
* Disease duration from the onset of multiple sclerosis symptoms less than (<) 15 years in participants with an EDSS score greater than (>) 5.0 at Screening
* Either treatment-naive or receiving treatment with disease-modifying therapies, including prior use of interferon (IFN)-beta-1a (Avonex®, Rebif®), IFN-beta-1b (Betaseron®/Betaferon), or glatiramer acetate (Copaxone®).
* At least one clinically documented relapse in the past year and/or at least one T1-weighted Gadolinium (Gd)-enhancing lesion in the past year and/or at least one new T2 lesion in the past year at the time of enrollment

Inclusion Criteria Specific to RMS Cohort Arm 4 Participants:

* Must meet inclusion criteria for the RMS cohort
* Separate signed Informed Consent Form for the RMS Delayed Time to Start Control Arm (Arm 4)
* Must be willing to remain on the same dose and regimen of current standard of care, or no treatment if treatment-naïve, for 12 weeks after study enrollment The treating and/or study physician must agree that the participant is eligible to remain on the same dose and regimen of their current standard of care at Screening, or to receive no treatment if the participant is treatment-naïve, for 12 weeks after study enrollment

Inclusion Criteria Specific to PPMS Participants:

* Diagnosis of PPMS in accordance with the 2010 revised McDonald criteria
* EDSS score of 3.0 - 6.5 points, inclusive, at Screening
* Disease duration from the onset of multiple sclerosis symptoms <10 years in participants with an EDSS at Screening less than or equal to (</=) 5.0
* Documented history of either elevated immunoglobulin G (IgG) Index or one or more IgG oligoclonal bands (OCBs) detected by isoelectric focusing

Exclusion Criteria:

* Diagnosis of secondary progressive multiple sclerosis without relapses for at least 1 year
* History or known presence of recurrent or chronic infection (e.g., human immunodeficiency virus [HIV], syphilis, tuberculosis)
* History of recurrent aspiration pneumonia requiring antibiotic therapy
* History of cancer, including solid tumors and hematological malignancies (except basal cell, in situ squamous cell carcinomas of the skin, and in situ carcinoma of the cervix of the uterus that have been excised and resolved with documented clean margins on pathology)
* History of or currently active primary or secondary immunodeficiency
* History of coagulation disorders
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* History of alcohol or other drug abuse within 24 weeks prior to enrollment
* Known presence or history of other neurologic disorders Significant, uncontrolled disease, such as cardiovascular (including cardiac arrhythmia), pulmonary (including chronic obstructive pulmonary disease), renal, hepatic, endocrine, gastrointestinal, or any other significant disease
* Congestive heart failure (according to New York Heart Association III or IV functional severity)
* Known active bacterial, viral, fungal, mycobacterial infection, or any major episode of infection requiring hospitalization or treatment with IV antibiotics
* Any concomitant disease that may require chronic treatment with systemic corticosteroids or immunosuppressants during the course of the study
* Contraindications or intolerance to oral or IV corticosteroids, including IV methylprednisolone, according to the country label
* Contraindication for LP
* Previous treatment with B cell-targeted therapies (such as rituximab, ocrelizumab, atacicept, belimumab, or ofatumumab)
* Previous treatment with natalizumab/Tysabri®, alemtuzumab, anti-CD4 agents, cladribine, teriflunomide, cyclophosphamide, mitoxantrone, azathioprine, mycophenolate mofetil, cyclosporine, methotrexate, total body irradiation, or bone marrow transplantation
* Treatment with fingolimod/Gilenya®, dimethyl fumarate/Tecfidera®, or similar treatment within 6 months prior to enrollment
* Receipt of a live vaccine within 6 weeks prior to enrollment
* Systemic corticosteroid therapy within 4 weeks prior to Baseline
* Previous or concurrent treatment with any investigational agent or treatment with any experimental procedure for multiple sclerosis (such as treatment for chronic cerebrospinal venous insufficiency)
* Certain laboratory abnormalities or findings at Screening
* Inability to complete an MRI
* Lack of peripheral venous access
* Pregnant or lactating, or intending to become pregnant during the study

Exclusion Criteria Specific to RMS Participants:

* Diagnosis of PPMS or secondary progressive multiple sclerosis without relapses

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2016-04-29 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- United States (12):
  - Stanford University, Palo Alto, California
  - University of California at San Francisco, San Francisco, California
  - University Of Colorado, Aurora, Colorado
  - Yale University School of Medicine ; Pulmonary & Critical Care, New Haven, Connecticut
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Washington University; Wash Uni. Sch. Of Med, St Louis, Missouri
  - Empire Neurology, PC, Latham, New York
  - Weill Cornell MC-NY Presbyter; Dept. of Neurology/Neuroscience, Judith Jaffe Multiple Sclerosis Ctr, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Ohio State University, Columbus, Ohio
  - Oklahoma Medical Research Foundation; MS Center of Excellence, Oklahoma City, Oklahoma
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Canada (2):
  - University of British Columbia Hospital Site; Djavad Mowafaghian Centre for Brain Health, Vancouver, British Columbia
  - McGill University; Montreal Neurological Institute; Neurological and Psychiatric, Montreal, Quebec
- Germany (2):
  - Universitätsklinikum "Carl Gustav Carus" der Technischen Universität Dresden, Dresden
  - Universitätsmedizin Göttingen Georg-August-Universität, Göttingen
- Karolinska Universitetssjukhuset, Solna, Stockholm, Sweden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 131 patients enrolled at 17 study locations in the U.S., Canada, Germany, and Sweden
Period: Overall Study
Arm/Group | RMS Cohort Arm 1: Ocrelizumab + LP | RMS Cohort Arm 2: Ocrelizumab + LP | RMS Cohort Arm 3: Ocrelizumab + LP | RMS Cohort Arm 4: Ocrelizumab + LP | PPMS Cohort: Ocrelizumab + LP
Started | 23 | 31 | 28 | 18 | 31
Completed | 0 | 0 | 0 | 0 | 1
Not Completed | 23 | 31 | 28 | 18 | 30
Not completed — Adverse Event | 1 | 2 | 2 | 0 | 0
Not completed — Continued Onto Commercially Available Ocrelizumab | 12 | 12 | 14 | 14 | 21
Not completed — Death | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 2 | 0 | 1 | 1 | 1
Not completed — Non-Compliance With Study Drug | 1 | 3 | 1 | 0 | 1
Not completed — Other | 3 | 4 | 1 | 0 | 0
Not completed — Physician Decision | 2 | 2 | 0 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 2 | 1 | 0
Not completed — Study Terminated By Sponsor | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 8 | 7 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RMS Cohort Arm 1: Ocrelizumab + LP | RMS Cohort Arm 2: Ocrelizumab + LP | RMS Cohort Arm 3: Ocrelizumab + LP | RMS Cohort Arm 4: Ocrelizumab + LP | PPMS Cohort: Ocrelizumab + LP | Total
Number analyzed (Participants) | 23 | 31 | 28 | 18 | 31 | 131
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 31 | 28 | 18 | 31 | 131
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.0 (10.4) | 38.7 (10.4) | 34.6 (10.8) | 36.4 (9.8) | 44.9 (7.4) | 38.5 (10.4)
Sex/Gender, Customized [Number; unit: Participants]
  Male | 8 | 9 | 8 | 7 | 16 | 48
  Female | 15 | 22 | 20 | 11 | 15 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 0 | 2 | 6
  Not Hispanic or Latino | 22 | 28 | 27 | 17 | 28 | 122
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 1 | 3 | 0 | 9
  White | 21 | 28 | 25 | 13 | 29 | 116
  More than one race | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Levels of NfL (Neurofilament Light) in CSF From Treatment Baseline to Post-Treatment With Ocrelizumab
Description: Primary Analysis was based on following data-cut off:
  Arm 1: Baseline to post-treatment at 12 weeks Arm 2: Baseline to post-treatment at 24 weeks Arm 3: Baseline to post-treatment at 52 weeks Arm 4: Baseline to post-treatment at 12 weeks PPMS Cohort: Baseline to post-treatment at 52 weeks
Time Frame: From Baseline to post-treatment (Week 12, 24, 52 according to randomization and Weeks 144 and 240)
Population: The ITT population is defined as all patients enrolled in the study who received at least one dose of Ocrevus
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | RMS Cohort Arm 1: Ocrelizumab + LP | RMS Cohort Arm 2: Ocrelizumab + LP | RMS Cohort Arm 3: Ocrelizumab + LP | RMS Cohort Arm 4: Ocrelizumab + LP | PPMS Cohort: Ocrelizumab + LP
Number analyzed (Participants) | 21 | 25 | 22 | 16 | 28
pg/mL
  Primary Analysis | -1232.97 (2060.37) | -1169.13 (1739.49) | -1008.13 (1132.68) | -931.83 (2816.27) | 261.85 (1175.72)
  LTE phase Week 144 | -2331.89 (3334.80) | -644.50 (1371.39) | -1287.58 (1822.72) | -2544.33 (3807.94) | -925.32 (2507.97)
  LTE phase Week 240 | -2499.98 (3606.71) | -791.51 (1150.89) | -1060.33 (1678.95) | -5488.70 (4350.46) | -1221.33 (2738.19)

2. Primary Outcome: Change in Number of CD19+ B Cells in CSF From Treatment Baseline to Post-Treatment With Ocrelizumab
Description: Arm 1: Baseline to post-treatment at 12 weeks Arm 2: Baseline to post-treatment at 24 weeks Arm 3: Baseline to post-treatment at 52 weeks Arm 4: Baseline to post-treatment at 12 weeks PPMS Cohort: Baseline to post-treatment at 52 weeks
Time Frame: From Baseline to post-treatment (Week 12, 24, 52 according to randomization and Weeks 144 and 240)
Population: The ITT population is defined as all patients enrolled in the study who received at least one dose of Ocrevus
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | RMS Cohort Arm 1: Ocrelizumab + LP | RMS Cohort Arm 2: Ocrelizumab + LP | RMS Cohort Arm 3: Ocrelizumab + LP | RMS Cohort Arm 4: Ocrelizumab + LP | PPMS Cohort: Ocrelizumab + LP
Number analyzed (Participants) | 21 | 25 | 22 | 16 | 28
cells/μL
  Primary Analysis | -0.22 (0.26) | -0.15 (0.36) | -0.13 (0.32) | -0.18 (0.37) | -0.09 (0.11)
  LTE phase Week 144 | -0.11 (0.08) | -0.14 (0.20) | -0.06 (0.23) | 0.15 (0.10) | -0.01 (0.09)
  LTE phase Week 240 | -0.08 (0.09) | -0.20 (0.26) | -0.02 (0.01) | -0.04 (0.05) | 0.01 (0.03)

3. Primary Outcome: Change From Baseline in Number of CD3+ T-Cells in CSF Post-Treatment With Ocrelizumab
Description: as for outcome 2
Time Frame: From Baseline to post-treatment (Week 12, 24, 52 according to randomization and Weeks 144 and 240)
Population: The ITT population is defined as all patients enrolled in the study who received at least one dose of Ocrevus
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | RMS Cohort Arm 1: Ocrelizumab + LP | RMS Cohort Arm 2: Ocrelizumab + LP | RMS Cohort Arm 3: Ocrelizumab + LP | RMS Cohort Arm 4: Ocrelizumab + LP | PPMS Cohort: Ocrelizumab + LP
Number analyzed (Participants) | 21 | 25 | 22 | 16 | 28
cells/μL
  Primary Analysis | -6.61 (10.48) | -1.92 (3.15) | -1.46 (2.67) | -1.98 (5.10) | -3.25 (4.32)
  LTE phase Week 144 | -3.45 (2.33) | 1.78 (9.76) | -0.83 (4.64) | 2.25 (0.17) | -3.62 (5.56)
  LTE phase Week 240 | -3.00 (3.16) | -3.47 (2.31) | -1.41 (1.30) | -1.67 (2.42) | -1.37 (0.54)

ADVERSE EVENTS:
Time Frame: From baseline up to 5 years
Description: Safety population is defined as all enrolled patients who received at least one infusion of ocrelizumab, even if the infusion was incomplete.
Arm/Group | RMS Cohort Arm 1: Ocrelizumab + LP | RMS Cohort Arm 2: Ocrelizumab + LP | RMS Cohort Arm 3: Ocrelizumab + LP | RMS Cohort Arm 4: Ocrelizumab + LP | PPMS Cohort: Ocrelizumab + LP
All-Cause Mortality (participants affected / at risk) | 1/23 | 0/31 | 0/28 | 0/18 | 1/31
Serious Adverse Events (participants affected / at risk) | 5/23 | 5/31 | 1/28 | 5/18 | 9/31
Other Adverse Events (participants affected / at risk) | 23/23 | 28/31 | 27/28 | 17/18 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RMS Cohort Arm 1: Ocrelizumab + LP (N=23) | RMS Cohort Arm 2: Ocrelizumab + LP (N=31) | RMS Cohort Arm 3: Ocrelizumab + LP (N=28) | RMS Cohort Arm 4: Ocrelizumab + LP (N=18) | PPMS Cohort: Ocrelizumab + LP (N=31)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seronegative arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple sclerosis relapse (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myelitis transverse (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Assisted suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RMS Cohort Arm 1: Ocrelizumab + LP (N=23) | RMS Cohort Arm 2: Ocrelizumab + LP (N=31) | RMS Cohort Arm 3: Ocrelizumab + LP (N=28) | RMS Cohort Arm 4: Ocrelizumab + LP (N=18) | PPMS Cohort: Ocrelizumab + LP (N=31)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Palpitations (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Inner ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 1 (2)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (5) | 3 (3) | 2 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Facial pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2) | 3 (3) | 4 (8) | 5 (10)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 2 (4) | 1 (1) | 2 (6)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Pain (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Puncture site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 3 (4) | 1 (1) | 1 (1) | 2 (4)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 5 (5) | 2 (3) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 4 (4) | 2 (2) | 1 (1) | 4 (4) | 5 (5)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Ear infection (Infections and infestations) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Herpes zoster (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (3)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infected cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Nail bed infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (4) | 2 (2) | 5 (6)
Oral candidiasis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 4 (5) | 10 (13) | 4 (5) | 1 (1) | 2 (2)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (10) | 6 (12) | 10 (19) | 12 (28) | 13 (22)
Urinary tract infection (Infections and infestations) | 4 (5) | 5 (6) | 5 (9) | 7 (14) | 11 (41)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Chillblains (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 4 (5) | 2 (2) | 5 (9)
Infusion related reaction (Injury, poisoning and procedural complications) | 15 (36) | 9 (13) | 16 (32) | 11 (16) | 12 (38)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 2 (3) | 4 (5) | 4 (7) | 4 (4) | 6 (8)
Post procedural contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (2) | 2 (2) | 1 (2) | 0 (0) | 3 (3)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (4) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood iron decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza A virus test positive (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Occult blood (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 4 (5) | 2 (3) | 11 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 9 (10)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (5) | 1 (1) | 3 (4)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 4 (5)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 3 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (5) | 5 (6) | 3 (6) | 3 (7)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0) | 1 (3) | 1 (1) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Coordination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (3)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (4) | 6 (10) | 4 (4) | 4 (5) | 5 (5)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 1 (1) | 4 (4) | 2 (5) | 4 (6)
Lhermitte's sign (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple sclerosis pseudo relapse (Nervous system disorders) | 3 (5) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Muscle spasticity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Paraesthesia (Nervous system disorders) | 3 (4) | 2 (3) | 4 (5) | 2 (3) | 4 (7)
Restless arm syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sensory disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinus headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 5 (5)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnambulism (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Breast cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 8 (8)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (2) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 3 (5) | 1 (1) | 2 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-11-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT02688985/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-18): https://cdn.clinicaltrials.gov/large-docs/85/NCT02688985/SAP_001.pdf